CLINICAL TRIAL: NCT01156389
Title: Open-label, Randomised, Drug Interaction Study of Pyramax (Pyronaridine Artesunate) and the Protease Inhibitor Ritonavir in Healthy Volunteers
Brief Title: Pyronaridine Artesunate-Ritonavir Drug-drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-010-10
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Malaria
Keywords: malaria; artemisinin-based combination therapy (ACT); antimalarial; pyronaridine artesunate (Pyramax)
MeSH Terms: conditions — Malaria | interventions — Ritonavir; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A Ritonavir plus Pyramax (Active Comparator): 7 days of ritonavir followed by 3 days of ritonavir plus Pyramax followed by 7 days of ritonavir followed by a 33 day follow-up period (40 days since last Pyramax dosing) and a study completion evaluation.
  Interventions: Drug: Ritonavir and Pyramax
- Arm B Pyramax (Active Comparator): 3 day treatment course of Pyramax, followed by a follow up period of 40 days since last Pyramax dosing and a study completion evaluation.
  Interventions: Drug: Pyramax

INTERVENTIONS:
Drug: Ritonavir and Pyramax — 100 mg ritonavir (one soft gelatin capsule twice per day over 17 days, the evening capsule on day 1 will be omitted) and Pyramax (pyronaridine/artesunate) 180:60 mg (3 to 4 tablets once per day according to weight for 3 days).
  Arms: Arm A Ritonavir plus Pyramax
Drug: Pyramax — Pyramax (pyronaridine/artesunate) 180:60 mg (3 to 4 tablets once per day according to weight for 3 days).
  Other Names: pyronaridine artesunate, PA
  Arms: Arm B Pyramax

SUMMARY:
The primary objective of the study is to determine any drug interaction between the antimalarial Pyramax (pyronaridine artesunate) and the protease inhibitor ritonavir in healthy subjects. The secondary objective of the study is to assess further the safety of Pyramax in this setting.

DETAILED DESCRIPTION:
This is a phase I, open label, randomized study to determine any drug interaction between Pyramax (pyronaridine/artesunate) and the protease inhibitor ritonavir in healthy volunteers. A total of 34 healthy volunteers (17 per treatment arm) will be enrolled in the study so that at least 30 (15 per treatment arm) will complete it. Subjects will be randomly assigned in a 1:1 ratio to receive either ritonavir (100 mg) twice daily for 17 days from Day 1-17 plus Pyramax (180:60 mg) once daily for 3 days from Day 8-10 in Arm A or pyronaridine/artesunate (180:60 mg) alone once daily for 3 days from Day 1-3 in Arm B.

Subjects will come to the clinic the evening before first dosing of Pyramax / ritonavir. If enrolled, and according to the treatment arm, subjects will stay in the clinic and attend subsequent visits as follows:

Arm A:

* Inpatient day -1 (evening) to day 17
* Ambulatory clinic visit once daily (morning) on day 22, 29, 36, 43 and 50 (end of study visit)

Arm B:

* Inpatient day -1 (evening) to day 4 (morning),
* Ambulatory clinic visit once daily (morning) on Day 5, 6, 8, 15, 22, 29, 36, and 43.(end of study visit) The subjects will be evaluated for pharmacokinetic parameters and safety/tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18 and 55 years with a body weight between 50 and 90 kg and a body mass index calculated using Quetelet's Index - weight (kg)/height (m2) between 18.5-30.0
2. Signed and dated a written informed consent form (ICF) before undergoing any study related activities, including discontinuation of any prohibited medications
3. Medically normal subjects with no significant abnormal findings at the screening physical examination as evaluated by the investigator
4. Strictly normal values of ALT, AST and bilirubin and normal or abnormal and clinically insignificant results (if agreed by the Investigator and the Sponsor on a case by case evaluation) of the other blood and urine laboratory parameters at screening
5. Female subjects of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who was post-menopausal (i.e., one year without menses) or who has undergone sterilization (via hysterectomy or bilateral tubal ligation)
6. Female subjects of childbearing potential with a negative urine pregnancy test at screening and a negative plasma pregnancy test prior to inclusion and who agreed to one of the following methods:

   * Double barrier method of contraception for 2 weeks before first study drug administration and throughout the entire study follow up period
   * Partner(s) who had undergone vasectomy and has been negative for sperm for at least 6 months
7. The ability to understand the requirements of the study and willingness to comply with all study procedures

Exclusion Criteria:

1. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, acute QTc interval greater or equal to 450 mseconds), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other clinical abnormality
2. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine or artesunate or other artemisinins or ritonavir
3. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
4. Seropositive HIV antibody
5. Previous participation in any clinical study with Pyramax
6. Presence or recent history (last two years) of tobacco abuse (≥10 cigarettes/day)
7. Known or suspected alcohol abuse or illicit drug use in the last 10 years before the study start or positive findings on urine drug screen
8. Intake of grapefruit and grapefruit juice alcoholic beverages or caffeine-containing food or beverages, such as coffee, tea, chocolate, or cola, 48 hours before study drug administration
9. Use of over-the-counter (OTC) medications, including vitamins, analgesics, or antacids, 1 week before the study start
10. Use of prescription medications 14 days before the study start or required chronic use of any prescription medication
11. Use of enzyme-altering agents (e.g., barbiturates, phenothiazines, cimetidine, etc.) within 30 days or 5 half lives, whichever the longer, before the study start
12. Plasma donation 1 month before the study start
13. Blood donation of 450 mL or more in the last 3 months before the study start
14. Participation in any clinical study in last 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Borghini Fuhrer, PhD, Study Director — Medicines for Malaria Venture
Locations (1):
- Covance Clinical Research Unit AG, Allschwil, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Ritonavir Plus Pyramax: 7 days of ritonavir followed by 3 days of ritonavir plus Pyramax followed by 7 days of ritonavir
- Arm B Pyramax: 3 day treatment course of Pyramax
Period: Overall Study
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax
Started | 17 | 17
Completed | 13 | 16
Not Completed | 4 | 1
Not completed — Elevated liver enzymes | 4 | 0
Not completed — Vomiting | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.6) | 43.7 (10.0) | 43.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 17 | 34
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (2.2) | 24.2 (2.6) | 23.65 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Analysis: Half-life, Tmax
Description: Half-life and Tmax for pyronaridine, artesunate, DHA:
  Tmax - time of the maximum observed concentration Half life - apparent plasma terminal elimination half-life, computed as ln (2)/Kel
  Blood samples for pyronaridine analysis were taken at Day 8 predose, Day 9 predose, Day 10 predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours postdose, and Days 11,12, 13, 15, 22, 29, 36 and 43.
  Blood samples for artesunate / DHA analysis were taken at Day 10 predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours postdose.
Time Frame: Until Day 50 for Arm A and until Day 43 for Arm B
Population: Number of subjects studied
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax
Number analyzed (Participants) | 17 | 17
hours
  Pyronaridine half- life (adjusted to a common dose of 9.72 mg/kg): number analyzed (Participants) | 15 | 16
  Pyronaridine half- life (adjusted to a common dose of 9.72 mg/kg) | 384 (223.2) | 321.6 (69.6)
  Pyronaridine Tmax (adjusted to a common dose of 9.72 mg/kg): number analyzed (Participants) | 17 | 16
  Pyronaridine Tmax (adjusted to a common dose of 9.72 mg/kg) | 2.32 (2.16) | 1.44 (0.36)
  Artesunate half-life (adjusted to common dose of 3.25 mg/kg): number analyzed (Participants) | 9 | 13
  Artesunate half-life (adjusted to common dose of 3.25 mg/kg) | 0.425 (0.131) | 0.465 (0.197)
  Artesunate Tmax (adjusted to common dose of 3.25 mg/kg): number analyzed (Participants) | 17 | 16
  Artesunate Tmax (adjusted to common dose of 3.25 mg/kg) | 1.22 (0.69) | 0.84 (0.43)
  DHA half-life (adjusted for common 3.25 mg/kg artesunate dose): number analyzed (Participants) | 16 | 14
  DHA half-life (adjusted for common 3.25 mg/kg artesunate dose) | 2.27 (1.04) | 2.35 (0.900)
  DHA Tmax (adjusted for common 3.25 mg/kg artesunate dose): number analyzed (Participants) | 17 | 16
  DHA Tmax (adjusted for common 3.25 mg/kg artesunate dose) | 1.90 (0.71) | 1.44 (0.403)

2. Primary Outcome: Pharmacokinetics Analysis: Cmax
Description: Cmax for pyronaridine, artesunate, DHA:
  Cmax - maximum peak observed concentration
  Blood samples for pyronaridine analysis were taken at Day 8 predose, Day 9 predose, Day 10 predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours postdose, and Days 11,12, 13, 15, 22, 29, 36 and 43.
  Blood samples for artesunate / DHA analysis were taken at Day 10 predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours postdose.
Time Frame: Until Day 50 for Arm A and until Day 43 for Arm B
Population: Number of subjects studied
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax
Number analyzed (Participants) | 17 | 17
ng/ml
  Pyronaridine Cmax (adjusted to a common dose of 9.72 mg/kg): number analyzed (Participants) | 17 | 16
  Pyronaridine Cmax (adjusted to a common dose of 9.72 mg/kg) | 480.2 (145.1) | 407.5 (167.1)
  Artesunate Cmax (adjusted to common dose of 3.25 mg/kg): number analyzed (Participants) | 17 | 16
  Artesunate Cmax (adjusted to common dose of 3.25 mg/kg) | 128.2 (91.2) | 108.7 (49.1)
  DHA Cmax (adjusted for common 3.25 mg/kg artesunate dose): number analyzed (Participants) | 17 | 16
  DHA Cmax (adjusted for common 3.25 mg/kg artesunate dose) | 611.4 (273.4) | 779.2 (267.5)

3. Secondary Outcome: Summary of Treatment Emergent Adverse Events
Description: Including all the treatment emergent adverse events, the number of subjects discontinued due to adverse events and the number of subjects with serious adverse events.
Time Frame: Throughout the study
Population: Number of subjects studied
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax
Number analyzed (Participants) | 17 | 17
Participants
  Mild treatment emergent adverse events | 12 | 15
  Moderate treatment emergent adverse events | 6 | 3
  Severe treatment emergent adverse events | 0 | 0
  Subjects discontinued due to adverse events | 4 | 1
  Subjects with serious adverse events | 0 | 0

4. Primary Outcome: Pharmacokinetics Analysis: AUC0-tau, AUC0-∞
Description: AUC0-tau, AUC0-∞ for pyronaridine, artesunate, DHA:
  AUC0-tau - area under the concentration-time curve from Hour 0 to the scheduled time of the next dose AUC0-∞ - area under the concentration-time curve from Hour 0 through the last quantifiable concentration time
  Blood samples for pyronaridine analysis were taken at Day 8 predose, Day 9 predose, Day 10 predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours postdose, and Days 11,12, 13, 15, 22, 29, 36 and 43.
  Blood samples for artesunate / DHA analysis were taken at Day 10 predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours postdose.
Time Frame: Until Day 50 for Arm A and until Day 43 for Arm B
Population: Number of subjects studied
Measure: Mean (Standard Deviation); unit: hours*ng/ml
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax
Number analyzed (Participants) | 17 | 17
hours*ng/ml
  Pyronaridine AUC0-tau (adjusted to a common dose of 9.72 mg/kg): number analyzed (Participants) | 16 | 16
  Pyronaridine AUC0-tau (adjusted to a common dose of 9.72 mg/kg) | 229 (82) | 222 (80)
  Pyronaridine AUC0-∞ (adjusted to a common dose of 9.72 mg/kg): number analyzed (Participants) | 15 | 16
  Pyronaridine AUC0-∞ (adjusted to a common dose of 9.72 mg/kg) | 1244 (292) | 1318 (481)
  Artesunate AUC0-tau (adjusted to common dose of 3.25 mg/kg): number analyzed (Participants) | 9 | 13
  Artesunate AUC0-tau (adjusted to common dose of 3.25 mg/kg) | 185.4 (105.6) | 150 (60)
  Artesunate AUC0-∞(adjusted to common dose of 3.25 mg/kg): number analyzed (Participants) | 9 | 13
  Artesunate AUC0-∞(adjusted to common dose of 3.25 mg/kg) | 185.4 (105.6) | 149 (60)
  DHA AUC0-tau (adjusted for common 3.25 mg/kg artesunate dose): number analyzed (Participants) | 16 | 14
  DHA AUC0-tau (adjusted for common 3.25 mg/kg artesunate dose) | 1308 (544) | 1978 (622)
  DHA AUC0-∞ (adjusted for common 3.25 mg/kg artesunate dose): number analyzed (Participants) | 16 | 14
  DHA AUC0-∞ (adjusted for common 3.25 mg/kg artesunate dose) | 1310 (545) | 1982 (628)

ADVERSE EVENTS:
Time Frame: up to Day 50 (end of study)
Description: The condition of each subject was monitored throughout the study. In addition, any signs and symptoms were observed and elicited at least once a day by open questioning, such as "How have you been feeling since you were last asked?". Subjects were also encouraged to report spontaneously any adverse events during the study.
Arm/Group | Arm A Ritonavir Plus Pyramax | Arm B Pyramax
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 10/17 | 13/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Ritonavir Plus Pyramax (N=17) | Arm B Pyramax (N=17)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 8 (9)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (5)
Fatigue (General disorders) | 2 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 5 (6)
Hot flush (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No